CLINICAL TRIAL: NCT02969668
Title: Effectiveness and Safety of Interferon-free Antiviral Regimens for the Treatment of Chronic Hepatitis C Virus Infection Among Opioid-substituted Patients
Brief Title: Interferon-free Antiviral Treatment of Chronic Hepatitis C Virus Infection Among Opioid-substituted Patients
Acronym: INFO
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Jens Reimer, Prof. Dr. med. Jens Reimer, MBA; Head of Centre for Interdisciplinary Addiction Research (CIAR), Hamburg University, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: AI444-366
Record Dates: First submitted 2016-06-05; First posted 2016-11-21 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C, Chronic; Opioid-Related Disorders
Keywords: opioid substitution treatment; interferon-free direct acting antivirals; hepatitis c therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks

SUMMARY:
The primary objective of study will be to evaluate the effectiveness of interferon-free direct acting antivirals (IFN-free DAAs) in the treatment of chronic hepatitis C virus (HCV) among patients in opioid-substitution treatment (OST). We hypothesize that rates of sustained virological response will be comparable to non-OST populations. Secondary objectives include the evaluation of safety data, patients' adherence and patient reported outcome measures like functioning (disability), satisfaction with the treatment, health status, general health perceptions and health-related quality of life.

DETAILED DESCRIPTION:
The new interferon-free antiviral regimens for the treatment of chronic hepatitis C (CHC) infections achieve impressive sustained virological response (SVR) rates beyond 90%, with shorter treatment duration and reduced side effects, irrespective of previous treatment history or presence of advanced liver diseases.

In Europe, the majority of HCV infections have been acquired and transmitted through injecting drug use - therefore, people who inject drugs (PWID) represent the majority of individuals with CHC infections in the Western industrialized cultures. There are excellent therapeutic options for those PWID who are in OST, as the frequent treatment provider-patient contact allows regular diagnoses, a continuing monitoring, and a sustainable management of HCV-infection among these patients. However, despite the growing evidence that patients in OST can successfully be treated for HCV, the treatment uptake among this predominant risk group is still very low. The current evidence from non-drug using populations only have a limited impact on the willingness of physicians providing opioid substitution treatment (OST), hepatologists and infectiologists to provide antiviral HCV treatment with IFN-free DAAs and on the willingness of OST patients to enter such treatment. Accordingly, data on the effectiveness and safety of antiviral HCV treatment regimens with IFN-free DAAs among this relevant patient group are urgently needed. The aim of this prospective cohort study is to assess the effectiveness, safety and patient reported outcome measures of IFN-free DAAs for the treatment of CHC among OST patients.

The primary objective of this open-label, observational, prospective cohort study will be to evaluate the effectiveness of IFN-free DAAs regimens for the treatment of chronic HCV-infection among OST patients in real life clinical settings.

Patients will be treated for chronic HCV with any kind of registered IFN-free DAA protocol and in accordance with the respective SmPC. This ensures that that dosing and schedule are supported by Phase I or later research. The study physician will make any medical decisions with regard to type of medication and doses. The individual treatment duration depends on the respective treatment protocol. The study physician is responsible for any medical decision and will document treatment dosage, treatment schedule, treatment duration and outcome.

Effectiveness is defined as sustained virological response at week 12 and week 24 after end of treatment (SVR12 and SVR24). SVR rates will be compared with the literature on non-substance using populations on the basis of two-sided 95% confidence intervals. The sample size calculation revealed, that 295 OST patients (HCV treatment naïve/Non-responder/Relapser) eligible for treatment with IFN-free DAAs (according to the summary of product (SmPC)) have to be included. To account for dropouts, we consider an over-recruitment of 10%, resulting in 325 patients to be recruited.

Secondary objectives include the collection of safety data during the treatment phase until SVR12, patients' adherence, and patient reported outcome measures like functioning (disability), satisfaction with the treatment, health status, general health perceptions and health-related quality of life.

All analyses - effectiveness and safety - will be conducted as intention-to-treat (ITT) as well as per protocol (PP) analyses. The ITT sample is defined as the number of patients starting treatment (first dose), whereas the PP sample includes only patients with complete data for SVR24.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* opioid dependence according to ICD-10
* admission to opioid substitution treatment for at least 3 months
* Chronic hepatitis C infection with genotype 1-6
* eligibility for antiviral HCV treatment with IFN-free DAAs according to the respective summary of product characteristics (SmPC)

Exclusion Criteria:

* missing eligibility for antiviral HCV treatment with IFN-free DAAs according to SmPC
* inability of the patient to participate in the study (e.g. due to severe mental impairment)
* missing patient-signed written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic HCV-genotype 1-6, aged over 18 years, who are for a minimum of 3 months in opioid substitution treatment and who are beginning an antiviral HCV treatment with interferon-free direct acting antivirals (IFN-free DAAs)
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2016-03; Primary Completion 2018-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | through study completion, up to 36 weeks after baseline
  Sustained virological response (SVR), defined as undetectable HCV RNA, will be assessed up to 36 weeks after baseline The individual treatment duration depends on the respective treatment protocol and varies between 8 and 24 weeks.

SECONDARY OUTCOMES:
Adverse events | through study completion, up to 36 weeks after baseline
  An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation subject administered study drug and that does not necessarily have a causal relationship with this treatment.
Patient-reported physical health status, as measured with the Opiate Treatment Index Health Scale (OTI-HSS) | through study completion, up to 36 weeks after baseline
  Patient-reported physical health status, as measured with the Opiate Treatment Index Health Scale (OTI-HSS)
Patient-reported mental health status, as measured with the brief symptom inventory 18 (BSI-18) | through study completion, up to 36 weeks after baseline
  Patient-reported mental health status, as measured with the brief symptom inventory 18 (BSI-18)
Health related quality of life, as measured with the short form 12 (SF-12, version 1) | through study completion, up to 36 weeks after baseline
  Health related quality of life, as measured with the short form 12 (SF-12, version 1)
Questionnaire on patient-reported fatigue and subjective cognitive impairments | through study completion, up to 36 weeks after baseline
  This is a self-developed questionnaire with 12 items (5 items on fatigue, and 7 items on subjective cognitive deficits), each item to be rated on a 5-point Likert-Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Reimer, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (18):
- Germany (18):
  - Praxiszentrum im Tal (PIT), Munich, Bavaria
  - Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH, Berlin
  - Praxisgemeinschaft Turmstraße, Berlin
  - Praxis Gabriele U. Bellmann/ Norbert E. Lyonn Fachärzte für Allgemeinmedizin, Berlin
  - Praxis Micus, Berlin
  - Praxiszentrum Kaiserdamm, Berlin
  - Praxis D. Höpner/M. H. Besson, Berlin
  - Gemeinschaftspraxis Dres. Tietje, Koc, Schulte, Bremen
  - Gemeinschaftspraxis Gotenring, Cologne
  - MainFachArzt, Frankfurt
  - Medizentrum Hamburg, Hamburg
  - Kompetenzzentrum für Suchtmedizin und Infektiologie, Hanover
  - Praxiszentrum Friedrichsplatz, Kassel
  - CIM GmbH Infektiologische Praxisgemeinschaft Busch/Christensen, Munich
  - Schwerpunktpraxis "Concept", Munich
  - Praxis Lebentrau, München
  - Dres. Ulmer, Frietsch, Müller, Roll, Stuttgart
  - PG Mauruschat/Weilbrenner, Wuppertal

IPD SHARING:
Plan to Share IPD: Undecided